CLINICAL TRIAL: NCT04100408
Title: Inherited Genetic Susceptibility in Langerhans Cell Histiocytosis (LCH)
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Other Study IDs: AEPI17N1
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Histiocytosis, Langerhans-Cell
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (biospecimen collection): LCH patients and their parents undergo collection of saliva or buccal mucosa samples for genetic mutational analysis. Germline DNA from saliva or buccal brushing will be sequenced, genotyped, and analyzed.
  Interventions: Other: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Other: Biospecimen Collection — Undergo saliva or buccal mucosa collection
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
The long-term goal is to define the mechanisms of pathogenesis underlying Langerhans cell histiocytosis (LCH). The overall objectives of the current study are to characterize the role of SMAD6 inherited genetic variation on LCH susceptibility and identify germline genomic regions associated with LCH somatic mutations. Building from preliminary data, the central hypotheses are: (1) causal genetic variants in SMAD6 underlie susceptibility to LCH, and (2) differences in LCH-related somatic activating mutations by race/ethnicity are related to Amerindian (i.e., Native American) genetic ancestry. The Central hypothesis will be tested by pursuing the specific aims.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To comprehensively characterize germline variants in SMAD6 and their association with LCH.

II. To identify novel germline variants associated with LCH.

III.To determine the role of genetic ancestry on LCH-related somatic mutations.

EXPLORATORY OBJECTIVES:

I. To integrate clinical and epidemiologic questionnaire data with genetic risk factor data from the Primary Aims to more comprehensively elucidate LCH susceptibility.

OUTLINE:

Case identification and recruitment followed by questionnaires and specimen processing.

ELIGIBILITY:
Inclusion Criteria:

* ≤ 25 years old at the time of original LCH diagnosis
* The patient must be enrolled on ACCRN07 and/or APEC14B1 and registered with COG by a North American member institution
* The patient must have a diagnosis of LCH (ICD Codes/Morphology: 9751/1; 9752/1; 9753/1; or 9754/3).
* The patient must be diagnosed with LCH on or after January 1, 2008.
* All questionnaire respondents must understand English or Spanish.
* All patients and/or their parents or legal guardians must provide informed consent.
* All institutional, FDA, and NCI requirements for human studies must be met.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with Langerhans cell histiocytosis (LCH) on or after January 1, 2008.
Sampling Method: Non-Probability Sample
Enrollment: 647 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Characterized germline variants in SMAD6 and their association with Langerhans Cell Histiocytosis (LCH) | Up to 4 years
  Will re-sequence SMAD6 among LCH case-parent trios to characterize the association between SMAD6 inherited genetic effects and LCH susceptibility using targeted next-generation sequencing. We will also analyze de novo single-nucleotide variants (SNVs), copy-number variants (CNVs), and insertions/deletions(INDELs) obtained through SMAD6 sequence data generated from the biologic samples of the CCRN/PEC LCH case-parent trios.
The frequency of de novo mutations and systematic assessment of the underlying genetic makeup of LCH | Up to 4 years
  Will use the maximum number of LCH case-parent trios enrolled utilizing the CCRN/PEC with viable biologic samples to conduct genome-wide SNP genotyping. This methodology will identify new genes and pathways associated with LCH susceptibility. We will also determine the prevalence of novel de novo mutations associated with LCH in these case-parent trios. This will provide a systematic assessment of the underlying genetic makeup of LCH in a large sample of families.
The difference in LCH-related somatic mutations by race/ethnicity due to underlying genetic ancestry | Up to 4 years
  Genetic ancestry will be determined using germline genome-wide SNP array data generated from CCRN/PEC LCH cases in Aim 2. In parallel, we will determine patient somatic mutational profiles using a custom, targeted 91-gene panel. We will then conduct a genome-wide admixture-mapping scan to identify LCH-related loci that are associated with specific LCH somatic mutational profiles.

OTHER OUTCOMES:
The role of genetic ancestry on LCH-related somatic mutations | Up to 4 years
  The analysis of data generated in this outcome measure will be primarily descriptive in nature. the objective will be to characterize LCH case-parent trios based on demographic, epidemiologic, and clinical characteristics. Findings from primary outcome measures findings will be validated and will assess if the frequency of validated inherited genetic variants differs by these characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Scheurer, PhD, Principal Investigator — Children's Oncology Group
Locations (1):
- Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas, United States